CLINICAL TRIAL: NCT07145424
Title: The Therapeutic Role of Kinesio Taping in Primary Dysmenorrhea: Reducing Pain and Enhancing Functionality: A Randomized Controlled Study
Brief Title: The Therapeutic Role of Kinesio Taping in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, özge ece günaydın, Assistant Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADU-FTR-EG-02
Record Dates: First submitted 2025-08-19; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Primary Dysmenorrhea; Pain Management
Keywords: dysmenorrhea; quality of life; rehabilitation; pain
MeSH Terms: conditions — Agnosia; Dysmenorrhea; Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were blinded to their group assignments. Outcome assessors were not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesio taping group (Experimental): kinesio taping was applied to the KT group taping was initiated during the participants' second menstrual cycle
  Interventions: Other: kinesio taping group
- control (No Intervention): This group only received assessments.

INTERVENTIONS:
Other: kinesio taping group — The original Kinesio Tape (Kinesio Tex Classic Tape) was used for taping by a physiotherapist with 15 years of experience in the field. The tape was cut into an I-shape and applied to the lower abdominal and lumbo-sacral regions where the participants experienced pain, 10 days prior to the anticipated start of menstruation (Figure 2). The tapes were renewed after four days. This procedure was performed three times and the total taping period was completed as 12 days. The tapes were removed on the third day of menstruation and all outcome measurements were performed again for the post intervention measurements
  Arms: kinesio taping group

SUMMARY:
Purpose: Dysmenorrhea is one of the most common causes of disability in women's health worldwide. It affects women's daily activities and negatively affects their social life. It increases healthcare costs and constitutes a significant burden for both women and society. Therefore, interventions to improve dysmenorrhea are needed. The aim of the study is to examine the effect of kinesio taping (KT) intervention on pain, muscle strength, functional disability, physical activity level, and quality of life.

Methods: Participants with primary dysmenorrhea were divided into kinesio taping (KT) and control (C) groups. The KT group underwent consecutive taping for 12 days starting from the premenstrual week. Trunk muscle strength evaluation, visual analogue scale (VAS), the pressure pain threshold, menstrual distress questionnaire (MDQ), SF-36 quality of life scale, Oswestry disability index (ODI), international physical activity questionnaire (IPAQ) were used as outcome measures.

DETAILED DESCRIPTION:
Dysmenorrhea is a prevalent and commonly experienced menstrual issue, characterized by pain that typically starts a day prior to menstruation and persists for 2-3 days, adversely impacting the individual's quality of life and hindering their ability to work and study . Dysmenorrhea can be categorized into two main types: primary and secondary. Primary dysmenorrhea refers to the occurrence of menstrual pain without any identifiable underlying anatomical or physiological abnormalities. In contrast, secondary dysmenorrhea is associated with an identifiable anatomical or physiological condition that contributes to the menstrual discomfort. Prior research has found the prevalence of dysmenorrhea among adolescent girls to be as high as 90.0%, while studies within the local context have reported a range of 34.0% to 89.6% . Given the high prevalence of dysmenorrhea, effective management strategies are crucial. Physiotherapy modalities are also among the non-pharmacological approaches frequently used to manage dysmenorrhea. These interventions include electrotherapy, massage, and taping techniques. The impact of kinesio taping on primary dysmenorrhea has been a subject of research. The Kinesio tape, which shares characteristics similar to human skin and is also breathable, smooth, hypoallergenic, able to remain affixed to the target tissue for 3-5 days, and does not impede movement . It is commonly used to reduce pain, modulate muscle function, influence joint positioning, enhance blood flow, and augment proprioceptive feedback . In a comparative analysis of the impacts of kinesio taping versus connective tissue massage interventions on pain and quality of life in individuals with primary dysmenorrhea, it is observed that despite a notable improvement in pain intensity and generally favorable outcomes associated with kinesio taping administered over three menstrual cycles, connective tissue massage demonstrates a more pronounced improvement. The levels of anxiety experienced by participants and their perceptions regarding menstruation were not influenced . In another study in premenstrual syndrome, the efficacy of kinesio taping and thermal application was analyzed by employing the Menstrual Distress Complaint List.The results demonstrated a significant improvement in symptomatic alleviation when these two methods were utilized together. Kinesio taping was recommended for use in premenstrual syndrome as an easy and non pharmacological application. In a separate study comparing the effects of kinesio taping and spiral taping on menstrual pain and premenstrual syndrome, participants underwent the intervention six times, specifically 14 days prior to the beginning of their menstrual cycle. The results revealed that kinesio taping was effective in menstrual pain, while spiral taping was effective in both menstrual pain and premenstrual syndrome. A comprehensive review of the current literature reveals a notable deficiency of empirical research exploring the effects of kinesio taping on primary dysmenorrhea, both within national boundaries and on an international scale. The most frequently evaluated parameters in these studies are pain intensity and menstrual complaint list, however, these studies fail to examine the influence of dysmenorrhea on functional status. Considering this identified gap, the present study aimed to evaluate the influence of Kinesio tape on dysmenorrhea by conducting supplementary assessments, including abdominal and lumbar muscle strength, the degree of functional disability, levels of physical activity, and quality of life metrics.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-30
* No hormonal contraception or intrauterine devices in the last 3 months
* Regular menstruation (every 21-35 days) for the last 6 months
* Pain score of 5 or more according to VAS.

Exclusion Criteria:

* Gynecological diseases
* Chronic systemic diseases
* Pregnancy or multiparousus
* Psychotherapeutic medications

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only females who are currently going through monthly menstruation cycles (21-35 days)
Enrollment: 36 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | from baseline to 4th week
  The Visual Analogue Scale (VAS) was used to evaluate the intensity of menstrual pain experienced by participants.It is a valid, reliable, and easily understandable scale that has been employed in research to assess the severity of primary dysmenorrhea. VAS is widely recognized as the most common quantitative measure for assessing the intensity of pain, where "0" represents no pain and "10" represents the most severe pain experienced .
Pressure pain threshold assessment | from baseline to 4th week
  Trigger points, whether active or latent, can contribute to increased muscle tension and subsequently lead to musculoskeletal pain. The pressure pain threshold at trigger points in the lumbar region was assessed using an analog algometer. Participants were instructed to indicate when they first experienced pain, and the corresponding pressure value was documented .
Muscle strength measurement | from baseline to 4th week
  A handheld dynamometer (Lafayette Instrument Company, Lafayette®, Lafayette, LA, USA) was used to evaluate the maximal muscle strength of the trunk muscles. This device represents a cost-effective and portable tool for assessing muscular strength, which is commonly employed in clinical settings due to its high reliability and validity relative to more sophisticated laboratory-based dynamometers. Participants were instructed to exert maximum muscle force against the fixed dynamometer held by the therapist, and their strength was measured. To assess trunk flexor strength, participants were positioned in supine with knees slightly bent, arms at their sides, and head in neutral. The dynamometer was placed on the midpoint of the sternum, and participants were asked to lift their scapulae from the floor. Trunk extensor strength was evaluated with participants in the prone position.

SECONDARY OUTCOMES:
Menstrual distress questionnaire (MDQ) | from baseline to 4th week
  The MDQ was used to evaluate participants' menstrual-related complaints and experiences during the premenstrual, menstrual and intermenstrual phases. This valid and reliable tool consists of a list of 47 symptoms divided into 8 sub-symptom groups: pain, water retention, autonomic reaction, negative affect, concentration, behavior change, arousal, and control. Complaints are scored on a 5-point scale from 0 (no symptoms) to 4 (very severe)
SF-36 quality of life scale | from baseline to 4th week
  The SF-36 instrument was employed to evaluate the quality of life. The last 4 weeks are taken into consideration in the assessment. This scale consists of 36 items that evaluate eight distinct dimensions: physical functioning, social functioning, role limitations due to physical concerns, role limitations due to emotional difficulties, mental health, energy/vitality, pain, and overall health perception. The subscales assess health on a scale of 0-100, with 0 indicating poor health status and 100 indicating good health status
Oswestry disability index | from baseline to 4th week
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools.For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. Interpretation of scores are;0% to 20% minimal disability,21%-40% moderate disability, 41%-60% severe disability, and above %60 means back pain impinges on all aspects of the patient's life.
International physical activity questionnaire (IPAQ) | From baseline to 4th week
  IPAQ was used to determine the physical activity levels of the participants. IPAQ is a validated and reliable instrument employed to gather valid and comparable data on physical activity levels based on individuals' self-reports of their daily physical activities. The questionnaire inquires about the time spent engaged in physical activities over the past 7 days. Individual's activity level is categorized as low, moderate, high.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No